CLINICAL TRIAL: NCT04396834
Title: Behavioral Mechanisms of Lorcaserin Treatment for Smoking Cessation
Brief Title: Mechanisms of Lorcaserin for Smoking Cessation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Medication removed from the U.S. market by the The Food and Drug Administration
Sponsor: The Mind Research Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 04619
Record Dates: First submitted 2020-02-03; First posted 2020-05-21 (Actual); Results first posted 2023-03-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Tobacco Use Disorder; Smoking Cessation
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — lorcaserin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lorcaserin first, then placebo (Experimental): Participants first receive lorcaserin (10 mg BID) for 7 days. After a washout period of 7 days, they then receive placebo tablets (BID) for 7 days.
  Interventions: Drug: Lorcaserin Oral Tablet
- Placebo first, then lorcaserin (Experimental): Participants first receive placebo (BID) for 7 days. After a washout period of 7 days, they then receive lorcaserin (10 mg BID) for 7 days.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Lorcaserin Oral Tablet — Lorcasering 10mg Oral Tablet (BID)
  Other Names: Belviq
  Arms: Lorcaserin first, then placebo
Drug: Placebo oral tablet — Placebo Oral Tablet (BID)
  Other Names: Placebo pill
  Arms: Placebo first, then lorcaserin

SUMMARY:
Identifying new medication options is critical for curbing the health burdens of cigarette smoking. Currently approved smoking cessation medications act on nicotinic receptors, and additional work is needed to identify medications with alternate pharmacological targets. Based on evidence that the serotonin system plays a role in nicotine consumption and relapse, this study will examine whether a selective serotonin medication alters smoking-related behaviors and responses to cigarette smoking under controlled conditions, informing its potential utility for smoking cessation.

DETAILED DESCRIPTION:
Tobacco use remains the foremost cause of preventable deaths in the U.S. and worldwide. Advancing new smoking cessation therapies, including those with novel pharmacological targets, is a critical public health priority. The serotonin (5-hydroxtytryptamine; 5-HT) system is broadly implicated in the regulation of reward- related behavior, including drug seeking, in part reflecting its modulatory role in dopamine (DA) function. Recent studies show that targeted manipulation of the serotonin 5-HT2C receptor alters drug-related behavior; in particular, 5-HT2C receptor agonists are shown to reduce nicotine intake and reinstatement. Of the selective 5-HT2C receptor agonists, lorcaserin has the best near-term potential for repurposing as a smoking cessation therapy, having been approved by the U.S. Food and Drug Administration for weight management.

Preclinical findings implicate several potential behavioral mechanisms by which 5-HT2C receptor agonists might reduce drug intake, including drug-specific processes (e.g., incentive salience of drug cues, self-administration, reinstatement) and drug-nonspecific behaviors (e.g., reductions in impulsivity). To date, potential mechanisms of 5-HT2C receptor agonists have not been characterized in human studies. Given emerging interest in lorcaserin as a novel smoking cessation therapy, further studies are needed to evaluate its efficacy profile, including studies to evaluate candidate treatment mechanisms. This human laboratory investigation will examine the effects of lorcaserin vs. placebo on relapse-related outcomes using a double-blind, within-subjects, crossover design. Impulsivity subdomains will also be examined as candidate mechanisms for medication effects. By evaluating an approved 5-HT2C agonist with emergent efficacy for smoking cessation, this project has near-term potential to inform clinical applications of 5-HT2C agonists for addiction.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-65
2. smoking 5+ cigarettes per day (average) over the past year, with no period of abstinence > 90 days
3. biochemical verification of smoking status
4. at least low to moderate nicotine dependence
5. reporting long-term motivation to quit smoking
6. willingness to take study pills and complete study procedures
7. willingness to complete lab sessions involving cigarette smoking

Exclusion Criteria:

1. meeting DSM-5 criteria for substance use disorder aside from tobacco use disorder and mild cannabis use disorder
2. recent (30 day) illicit drug use (except marijuana), based on self-report and urine drug screen
3. past 30-day use of tobacco cessation aids or nicotine/tobacco products other than cigarettes
4. past 30-day use of SSRIs, other psychiatric medications, or weight control medications
5. lifetime diagnosis of severe mental illness (e.g., psychotic or bipolar I disorder)
6. significant medical or neurological illness, including severe hepatic impairment or cirrhosis, or insulin dependent diabetes
7. actively engaged in smoking cessation treatments or a smoking cessation attempt (or intent to start an attempt in the next 90 days)
8. interested in quitting smoking immediately (i.e., in the next two months)
9. Medications contraindicated for use with lorcaserin or which have a significant interaction with lorcaserin
10. body mass index (BMI) under normal range (BMI < 18 kg/m2)
11. history of significant cardiovascular conditions including history of arrhythmias or heart block, heart failure, valvular heart disease, heart attack, stroke, unstable angina
12. abnormal electrocardiogram (ECG) results
13. nursing, pregnant, or anticipating pregnancy
14. history of suicide attempt or recent suicidal thoughts (intent or plan) in the last month
15. Plans to travel outside of the local area during the study period, or inability to commit to entire duration of study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 3 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Hendershot, Ph.D., Principal Investigator — The Mind Research Network; Eric Claus, Ph.D., Principal Investigator — The Mind Research Network
Locations (1):
- The Mind Research Network, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three participants provided informed consent. Due to the study being canceled, only two participants were assigned to condition.
Period: Overall Study
Arm/Group | Lorcaserin First, Then Placebo | Placebo First, Then Lorcaserin
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The trial was halted after randomizing the first two participants. Outcomes were not analyzed due to recruitment of only two participants.
Groups:
- Lorcaserin First, Then Placebo: Lorcaserin (10mg BID) for 7 days, then placebo pill (BID) for 7 days
- Placebo First, Then Lorcaserin: Placebo pill (BID) for 7 days, then lorcaserin (10mg BID) for 7 days
- Total: Total of all reporting groups
Arm/Group | Lorcaserin First, Then Placebo | Placebo First, Then Lorcaserin | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The trial was halted after randomizing the first two participants. Outcomes were not analyzed due to recruitment of only two participants.
  Participants
    Female | 1 | 0 | 1
    Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The trial was halted after randomizing the first two participants. Outcomes were not analyzed due to recruitment of only two participants.
  Participants
    Hispanic or Latino | 1 | 0 | 1
    Not Hispanic or Latino | 0 | 1 | 1
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The trial was halted after randomizing the first two participants. Outcomes were not analyzed due to recruitment of only two participants.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 1 | 1 | 2
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Population: The trial was halted after randomizing the first two participants. Outcomes were not analyzed due to recruitment of only two participants.
  Participants
    United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Smoking Lapse
Description: Duration (in minutes) until lapsing to smoking during a 50-minute period
Time Frame: Laboratory session following 7 days of medication or placebo pills
Population: The trial was halted after randomizing the first two participants.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Lorcaserin: Lorcaserin (10mg BID)
  Lorcaserin Oral Tablet: Lorcasering 10mg Oral Tablet (BID)
- Placebo: Placebo pill (BID)
  Placebo oral tablet: Placebo Oral Tablet (BID)
Arm/Group | Lorcaserin | Placebo
Number analyzed (Participants) | 2 | 2
minutes | 16.5 (4.9) | 30.5 (.71)

2. Primary Outcome: Laboratory Cigarette Smoking
Description: Number of cigarettes consumed during a 60-minute period
Time Frame: Laboratory session following 7 days of medication or placebo pills
Population: The trial was halted after randomizing the first two participants.
Measure: Mean (Standard Deviation); unit: number of cigarettes
Arm/Group | Lorcaserin | Placebo
Number analyzed (Participants) | 2 | 2
number of cigarettes | 4 (1.41) | 3 (1.41)

3. Secondary Outcome: Impulsivity
Description: Performance on a behavioral measure of impulsivity, the stop signal task. Reported is the stop signal reaction time, the number of milliseconds required to activate the "stop" process in the stop signal task.
Time Frame: Laboratory session following 7 days of medication or placebo pills.
Population: The trial was halted after randomizing the first two participants.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Lorcaserin | Placebo
Number analyzed (Participants) | 2 | 2
milliseconds | 280.2 (11.6) | 255.4 (34.5)

4. Secondary Outcome: Reward Sensitivity
Description: Performance on a behavioral measure of reward sensitivity (response bias measure on a signal detection task). Response bias is computed by the following equation: 1/2 * log((# correct stim 1 * # incorrect stim 2)/(# incorrect stim 1 * # correct stim 2))
  Stimulus 1 is associated with a higher proportion of correct feedback than Stimulus 2, and by computing the ratio above, we are able to determine the response bias of the participant. The response bias measure provides an objective measure of reward sensitivity (i.e., the degree to which participants are biased towards choosing the more frequently rewarded response).
Time Frame: Laboratory session following 7 days of medication or placebo pills.
Population: The trial was halted after randomizing the first two participants.
Measure: Mean (Standard Deviation); unit: log(ratio)
Arm/Group | Lorcaserin | Placebo
Number analyzed (Participants) | 2 | 2
log(ratio) | .89 (.51) | .80 (.41)

5. Secondary Outcome: Daily Cigarette Smoking
Description: Cigarettes smoked per day
Time Frame: During 7 days of medication or during 7 days of placebo pills (difference score between weeks).
Population: The trial was halted after randomizing the first two participants.
Measure: Mean (Standard Deviation); unit: cigarettes per day
Arm/Group | Lorcaserin | Placebo
Number analyzed (Participants) | 2 | 2
cigarettes per day | 8.79 (.30) | 8.79 (.30)

ADVERSE EVENTS:
Time Frame: 1 month
Groups:
- Lorcaserin: Lorcaserin (10mg BID) for 7 days
- Placebo: Placebo pill (BID) for 7 days
Arm/Group | Lorcaserin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 1/2 | 0/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lorcaserin (N=2) | Placebo (N=2)
Shingles (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Participant reported incident of shingles approximately one week following participation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-10): https://cdn.clinicaltrials.gov/large-docs/34/NCT04396834/Prot_SAP_000.pdf
  • Informed Consent Form (2019-09-10): https://cdn.clinicaltrials.gov/large-docs/34/NCT04396834/ICF_001.pdf